CLINICAL TRIAL: NCT06356766
Title: Investigation of Effectiveness of Modified Duran Protocol Via Telerehabilitation After Zone 2 Flexor Tendon Injury Repair of the Hand
Brief Title: Investigation of Effectiveness of Telerehabilitation for Zone 2 Flexor Tendon Injuries of the Hand
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fatma Merih Akpınar, Assistant Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30.01.2024/009
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Zone 2 Flexor Tendon Injuries of the Hand
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): Modified Duran Protocol via telerehabilitation
  Interventions: Other: Telerehabilitation
- Face-to-face Rehabilitation Group (Active Comparator): Modified Duran Protocol
  Interventions: Other: Face-to-face rehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Modified Duran Protocol via Telerehabilitation
  Arms: Telerehabilitation Group
Other: Face-to-face rehabilitation — Modified Duran Protocol
  Arms: Face-to-face Rehabilitation Group

SUMMARY:
The treatment process following Zone 2 flexor tendon injuries, which are particularly controversial for hand surgery, is challenging. There are various rehabilitation methods for Zone 2 flexor tendon injuries, one of which is the Modified Duran Protocol. Disruptions in the physiotherapy process lead to joint contractures, tendon adhesions, and limitations in daily life activities for patients. Due to global issues such as socioeconomic factors, physical barriers, distance, and pandemics, patients who cannot actively participate in physiotherapy miss out on the rehabilitation process.

The aim of the present study is to investigate the effectiveness of the Modified Duran protocol applied through telerehabilitation following Zone 2 flexor tendon repair. Between April and October 2024, a total of 42 adults aged 18-55 who underwent Zone 2 flexor tendon repair at Istanbul University Istanbul Faculty of Medicine will be recruited, with 21 participants in face-to-face clinic group and 21 in telerehabilitation group. Rehabilitation process will be followed for 12 weeks. The telerehabilitation group will receive exercise training on the third day. After the first training session, patients will be discharged and called to the clinic once a week for dressing changes, monitoring, exercises and if necessary, revision of the protective splint. Patients will be contacted three times a week to implement the planned program using telerehabilitation.

The face-to-face rehabilitation group will receive face-to-face clinic rehabilitation three times a week under the supervision of a physiotherapist for the first 12 weeks.

Patients will be evaluated at the end of the 5th, 6th, and 12th weeks. Data collection tools will include a 'Sociodemographic Form', 'Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire', 'Visual Analog Scale (VAS)', 'Jamar Hand Dynamometer', and 'Goniometer (Joint Range of Motion)'.

SPSS (Statistical Package for the Social Sciences) Statistics will be used for the statistical analysis of all data, with a significance level of p <0.05 considered significant in all assessments, and accepted as two-tailed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with isolated Zone 2 flexor digitorum profundus (FDP) and flexor digitorum superficialis (FDS) injuries,
* Repair performed within the first 72 hours post-injury,
* Individuals aged between 18 and 55 years,
* Patients willing to participate in the study,
* Ability to attend sessions regularly.

Exclusion Criteria:

* Fingers with concomitant fractures, digital nerve injuries, vascular injuries, or significant skin loss accompanying flexor tendon injuries,
* Bilateral flexor tendon injuries,
* Patients with replantation or revascularization,
* Flexor Pollicis Longus tendon injuries of the thumb due to differences in protocols applied and measurement of final outcomes,
* Patients unable to understand and perform postoperative exercises

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-11-08 (Estimated); Study Completion 2025-05-08 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | First week, 5th week, 6th week, 12th week
  Modified Strickland Formula

SECONDARY OUTCOMES:
DASH | First week, 5th week, 6th week, 12th week
  Disabilities of the Arm, Shoulder and Hand; min: 0 max: 100, lower scores indicate a lower level of disability
Pain of the affected hand | First week, 5th week, 6th week, 12th week
  Visual Analogue Scale, min:0 cm/mm, max: 10 cm/100 mm, higher scores mean a higher degree of pain
Muscle Strength | 12th week
  Jamar Hydraulic Hand Dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Seda Saka, Study Chair — Halic University
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No